CLINICAL TRIAL: NCT06100120
Title: A Triple-blinded Non-inferiority Multicentre Randomized Controlled Trial Comparing Hybrid and Fully Etched Implants.Part 1. Implant Stability.
Brief Title: A Triple-blinded Non-inferiority Multicentre Randomized Controlled Trial Comparing Hybrid and Fully Etched Implants P1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Giulio Rasperini, Associate Professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RCT Hybrid vs Fully etched P1
Record Dates: First submitted 2023-10-16; First posted 2023-10-25 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Dental Implants
Keywords: Implant stability; Implant surface; Hybrid Implants

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid implants (Experimental): Hybrid implants will be placed in this group
  Interventions: Procedure: Implant placement
- Fully etched implants (Active Comparator): Fully etched implants will be placed in this group
  Interventions: Procedure: Implant placement

INTERVENTIONS:
Procedure: Implant placement — Placement of osteointegrated implants

SUMMARY:
The goal of this randomized controlled clinical trial is to compare implant stability between hybrid implants and fully rough implants in partially edentulous patients. The main question it aims to answer is: are hybrid implants able to achieve a sufficient level of secondary stability in comparison to fully etched implants? Participants will receive dental implants and the secondary stability will be measured using resonance frequency analysis (RFA) at the 2-month post-implant placement mark. Implants that do not attain adequate secondary stability will undergo re-evaluation at monthly intervals up to 6 months. Researchers will compare the test group (hybrid implants) or the control group (fully rough implants) to see if they present a comparable secondary stability.

DETAILED DESCRIPTION:
This is a randomized triple-blinded, parallel-arm (1:1) controlled clinical trial with 6 months follow-up. Implants will be placed in 16 private practices. 128 patients will be randomly allocated to the test (hybrid implants)(64) and control (fully etched implants)(64) groups following stratified randomization in such a way that an equal number of patients in the test and in the control group will be enrolled in each study centre. The following individuals will be blinded as follows: 1) patients involved in the study will not be aware of the implants that are receiving; 2) surgeons: after the screening examination clinicians will choose the implant dimension but they will not be aware of the surface characteristic of the implant they are going to place until the implant socket is prepared; 3) the data collector/outcome assessor: of the implant stability will not be aware of the group allocation; 4) the statistician will not be aware of the group allocation. Treatment allocation will be concealed by using opaque sealed boxes and opened immediately before the implant placement (after implant socket preparation). At least 2 hours before the surgery all patients will be given antibiotic prophylaxis of 2g of amoxicillin (600mg of clindamycin for patients that allergic to penicillin). All implants (more than one implant per patient might be included) will be placed by 16 experienced surgeons in their respective clinic following according to the instruction provided by the manufacturer. The apicocoronal position of the implants will be equicrestal (i.e. the most coronal part of the machined collar is at the level of the alveolar ridge) or subcrestal (≤1 mm). In the test group and control group hybrid implants and fully etched implants (Volution, IRES®, Switzerland) will be placed. After surgery, in order to control discomfort and swelling, 600 mg ibuprofen every 8 hours if needed will be given. All subjects will be prescribed 0.12% chlorhexidine mouth rinse twice daily for 7 days. Immediately after the implant placement (Tpl) and at two months (T2) the implant stability will be measured using magnetic RFA (OsstellTM Mentor AB, Gothenburg, Sweden) by a trained clinician not involved in the study. The transducer will be screwed manually and RFA measurement were made both in the mesio-distal (MD) and bucco-lingual (BL) direction by keeping the device perpendicular at a distance between 2-4 mm and at least 3mm far away from the soft tissues. The peak insertion torque will be also registered. All implants will be submerged. Implants with ISQ values < 60 at the revaluation (T2) will undergo further measurements after 1 month till the 6th month after their placement. If at any timepoint (T2, T3, T4, T5, T6) the implant reaches a sufficient (stability ≥60) it will be considered stable till the end of the study, hence, no further ISQ assessment will be carried out and the prosthesis will be delivered (TL).

Continuous variables will be expressed as mean and standard deviation, whereas the absolute and relative frequency will be calculated for categorical variables. Regarding continuous variables, differences between groups will be tested by parametric or non-parametric test after testing the normal distribution of the data (Shapiro-Wilk test). For categorical variables chi-squared test (or Fisher test) will be adopted.

ELIGIBILITY:
Inclusion Criteria:

* Partially edentulous patients who need at least one fixed partial denture supported by 1 or 2 implants;
* Men and women over 20 years old;
* Periodontally stable patients
* Sufficient 3D bone availability
* Ideal 3D implant placement: MD: minimum tooth-implant distance of 1.5 mm and minimum inter-implant distance of 3 mm; at least 1.5 mm of buccal plate thickness; the implants should be placed equicrestally or 1 mm subcrestally in such a way that the machined part remains completely submerged; the distance between the implant neck and the adjacent dentition should be less than 6mm; straight implants (0 to 20 degrees from the adjacent tooth long axis or 70 to 90 degrees from the ridge parallelism);

Exclusion Criteria:

* Pregnant or lactating women;
* Uncontrolled systemic conditions;
* Patients on drugs known to interfere with the bone metabolism;
* Current smokers;
* Simultaneous/staged regenerative procedures;
* Immediate loading;
* Immediate implants;
* Short implants (< 8 mm) or narrow implant (diameter <3.3 mm);

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Secondary implant stability | 2 months, 3 months, 4 months, 5 months, 6 months
  Cumulative percentage of implants that achieve a successful secondary stability (ISQ>=60)

SECONDARY OUTCOMES:
Insertion torque | Day 0 (implant placement)
  Peak insertion torque measured during implant placement
Implant survival rate | 2 months, 3 months, 4 months, 5 months, 6 months
  Implants still present at each time point
Marginal bone level | Day 0, Day of prosthesis delivery
  Distance between implant shoulder and bone crest (mesial and distal)

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Rasperini, DDS, Principal Investigator — University of Milan
Locations (1):
- Clinica Odontoiatrica IRCCS Ospedale Maggiore Policlinico, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodrigo D, Aracil L, Martin C, Sanz M. Diagnosis of implant stability and its impact on implant survival: a prospective case series study. Clin Oral Implants Res. 2010 Mar;21(3):255-61. doi: 10.1111/j.1600-0501.2009.01820.x. Epub 2009 Dec 4. PMID 19958375
- [Background] Spinato S, Bernardello F, Sassatelli P, Zaffe D. Hybrid Implants in Healthy and Periodontally Compromised Patients: A Preliminary Clinical and Radiographic Study. Int J Periodontics Restorative Dent. 2017 Mar/Apr;37(2):195-202. doi: 10.11607/prd.3140. PMID 28196158
- [Background] Morton D, Gallucci G, Lin WS, Pjetursson B, Polido W, Roehling S, Sailer I, Aghaloo T, Albera H, Bohner L, Braut V, Buser D, Chen S, Dawson A, Eckert S, Gahlert M, Hamilton A, Jaffin R, Jarry C, Karayazgan B, Laine J, Martin W, Rahman L, Schlegel A, Shiota M, Stilwell C, Vorster C, Zembic A, Zhou W. Group 2 ITI Consensus Report: Prosthodontics and implant dentistry. Clin Oral Implants Res. 2018 Oct;29 Suppl 16:215-223. doi: 10.1111/clr.13298. PMID 30328196
- [Background] Berglundh T, Gotfredsen K, Zitzmann NU, Lang NP, Lindhe J. Spontaneous progression of ligature induced peri-implantitis at implants with different surface roughness: an experimental study in dogs. Clin Oral Implants Res. 2007 Oct;18(5):655-61. doi: 10.1111/j.1600-0501.2007.01397.x. Epub 2007 Jun 30. PMID 17608738
- [Background] Sennerby L, Meredith N. Implant stability measurements using resonance frequency analysis: biological and biomechanical aspects and clinical implications. Periodontol 2000. 2008;47:51-66. doi: 10.1111/j.1600-0757.2008.00267.x. No abstract available. PMID 18412573